CLINICAL TRIAL: NCT02780414
Title: Collection of Samples From Pregnant Women for the Evaluation of Preeclampsia (Pre-E) Biomarkers
Status: Completed | Type: Observational
Sponsor: Progenity, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-104-PREECLAMPSIA
Record Dates: First submitted 2016-05-12; First posted 2016-05-23 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Preeclampsia; Hypertension; Proteinuria; Thrombocytopenia; Renal Insufficiency; Impaired Liver Function; Pulmonary Edema
Keywords: Hypertension; Proteinuria; Thrombocytopenia; Renal Insufficiency; Impaired Liver Function; Pulmonary Edema
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Proteinuria; Thrombocytopenia; Renal Insufficiency; Liver Diseases; Pulmonary Edema

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This research study will collect 20 mL of whole blood and a 5 mL urine sample at one or more clinic visits from pregnant women carrying a single fetus with no known fetal abnormalities.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study Cohort: A group of at least 1,541 pregnant women with NO Pre-E diagnosis
- Positive Pre-E Control: A group of at least 250 pregnant women diagnosed with Pre-E

SUMMARY:
Preeclampsia (Pre-E) is a hypertensive disease of pregnancy with multi-system involvement that usually occurs in the second half of pregnancy. Pre-E occurs in 5% to 7% of U.S. pregnancies, and is the third-leading cause of U.S. maternal death. Improvements to the current diagnostic paradigm have been evaluated. However, no stand-alone diagnostic method has emerged that more accurately identifies women at risk for preeclampsia, warranting improvements in diagnosing Pre-E.

This sample collection study will obtain serum and urine samples from pregnant women who present with clinical signs, symptoms, or conditions contributing to the suspicion of Pre-E. Samples will be used to evaluate and validate the performance of an assay intended to aid in assessing the risk of Pre-E.

DETAILED DESCRIPTION:
Eligible subjects will provide written informed consent after which demographic and baseline clinical data will be recorded.

Collection of whole blood and urine samples will be performed at one or more clinic visits from pregnant women carrying a single fetus with no known fetal abnormalities.

Interim study visits will continue every 14 days [+/- 3 days] until the subject either: 1) reaches 37 0/7 weeks' gestation, 2) develops Pre-E, 3) delivers, or 4) is lost to follow-up.

In addition, a group of pregnant women diagnosed with Pre-E will be enrolled as positive control cases.

ELIGIBILITY:
Eligibility criteria for the STUDY COHORT (CASES and NEGATIVE PRE-E

CONTROLS):

Inclusion Criteria:

* Subject is willing to provide informed consent and comply with study procedures
* 18 to 45 years of age
* Singleton fetus of 28 0/7 to 36 6/7 weeks' gestational age using the 2014 American Congress of Obstetricians and Gynecologists (ACOG) Dating Criteria (pregnancies starting as twins but complicated with either vanishing twin syndrome or fetal demise of one twin before 14 weeks, are eligible for inclusion)
* Patient presenting with clinical suspicion of Pre-E based on either: New onset elevated blood pressure in otherwise normotensive patient, worsening hypertension in a patient with pre-existing hypertension, new onset proteinuria or worsening of pre-existing proteinuria, or any other clinical finding requiring a workup to rule-out Pre-E.

Exclusion Criteria:

* Pregnancy is non-viable or absence of fetal cardiac activity
* Diagnosis of Pre-E or anticipated delivery within 24 to 48 hours because of Pre-E with severe features including: persistent severe hypertension (systolic ≥160 or diastolic ≥110; thrombocytopenia <100,000; liver enzymes 2x above upper normal limit or >70 with severe persistent right upper quadrant (RUQ) or epigastric pain, new development of renal insufficiency; pulmonary edema; new-onset persistent cerebral or visual disturbances.
* Major fetal anomaly or chromosomal aneuploidy
* Current dialysis for kidney failure, including continuous ambulatory peritoneal dialysis

Eligibility criteria for the POSITIVE CONTROL group:

Inclusion Criteria:

* Subject is willing to provide informed consent and comply with study procedures
* 18 to 45 years of age
* Singleton fetus of 28 0/7 to 36 6/7 weeks' gestational age using 2014 ACOG Dating Criteria (pregnancies starting as twins but complicated with either vanishing twin syndrome or fetal demise of one twin before 14 weeks, are eligible for inclusion)
* Patient diagnosed with Pre-E using 2013 ACOG guidelines

Exclusion Criteria:

* Pregnancy is non-viable or absence of cardiac activity
* Major fetal anomaly or chromosomal aneuploidy
* Current dialysis for kidney failure, including continuous ambulatory peritoneal dialysis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women 18 to 45 years of age and 28 0/7 to 36 6/7 weeks gestational age with a singleton fetus presenting to clinic/triage/Labor & Delivery for evaluation of, but not limited to, one or more of the following:
  * new onset elevated blood pressure
  * pre-existing hypertension
  * new onset proteinuria or worsening of pre-existing proteinuria
  * other organ system findings including thrombocytopenia, renal insufficiency, impaired liver function, pulmonary edema, and cerebral or visual symptoms
Sampling Method: Non-Probability Sample
Enrollment: 1730 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Suspected and Pre-E cases determined by institutional standards | about 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stiegler, PhD, Study Director — Progenity, Inc.
Locations (20):
- United States (20):
  - Center of Research in Women's Health, Birmingham, Alabama
  - University of Colorado, Aurora, Colorado
  - Yale Medical, New Haven, Connecticut
  - Northwestern, Chicago, Illinois
  - Indiana University Health Physicians Women's Health, Indianapolis, Indiana
  - Johns Hopkins Medicine, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington Univ School of Medicine - Dept of OB-GYN, St Louis, Missouri
  - Winthrop Clinical Trials Center, Mineola, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Regional Obstetrical Consultants, PC, Chattanooga, Tennessee
  - Austin Maternal Fetal Medicine, Austin, Texas
  - University of Texas Medical Branch, Galveston, Galveston, Texas
  - UT Health Medical School, Houston, Texas
  - University of Utah Hospital, OB/GYN Dept., Salt Lake City, Utah
  - Medical College of Wisconsin - Department of Obstetrics & Gynecology, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Costantine MM, Sibai B, Bombard AT, Sarno M, West H, Haas DM, Tita AT, Paidas MJ, Clark EAS, Boggess K, Grotegut C, Grobman W, Su EJ, Burd I, Saade G, Chavez MR, Paglia MJ, Merriam A, Torres C, Habli M, Macones G, Wen T, Bofill J, Palatnik A, Edwards RK, Haeri S, Oberoi P, Mazloom A, Cooper M, Lockton S, Hankins GD. Performance of a Multianalyte 'Rule-Out' Assay in Pregnant Individuals With Suspected Preeclampsia. Hypertension. 2022 Jul;79(7):1515-1524. doi: 10.1161/HYPERTENSIONAHA.122.19038. Epub 2022 May 12. PMID 35545947